CLINICAL TRIAL: NCT01240369
Title: Association Between VEGF-C and miRNA and Clinical Non-small Cell Lung Cancer and Esophagus Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Jen-Liang Su, China Medical University Hospital
Other Study IDs: DMR99-IRB-206
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: VEGFC Protein in Serum; VEGFC Protein in Non Small Cell Lung Cancer; VEGFC Protein in ESCC; CTTN Protein in ESCC; miR326 in ESCC and Non Small Cell Lung Cancer
Keywords: VEGFC; CTTN; miR326; ESCC; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- VEGF-C low
- VEGF-C high
- miR-326 low
- miR-326 high

SUMMARY:
Lung cancer and esophageal cancer remain the leading causes of cancer death worldwide. The main problem is lack of effective tool in early detection that accounts for the poor outcome of cancer. Clinically, over 80% of patients with cancer were at late stage when they were diagnosed. Therefore, it is important for us to find the biomarker that serve as the early prediction of cancer.

The investigators have published that VEGFC over-expressed in non-small cell lung cancer. VEGFC plays a critical role in regulating motility of tumor cells, promotes proliferation of lymphatic endothelial cells and enhances migration and invasion. Investigator found that VEGFC over-expressed in the serum of esophageal cancer patients. Therefore, it is worthwhile to investigate the correlation between VEGFC, clinical lung cancer and esophageal cancer.

MicroRNAs (miRNAs) are conserved, endogenous, small, and noncoding RNA molecules of 21~23 nucleotides that function as post-transcriptional gene regulators. Recent studies indicated that certain microRNAs reduced in cancer patients. Therefore it is important to investigate whether specific microRNA changed in certain kinds of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* tumor size > 0.5 cm3

Exclusion Criteria:

* tumor size < 0.5 cm3

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESCC and NSCLC patients
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-10